CLINICAL TRIAL: NCT04759599
Title: Which is Better: Narrow vs. Wide Focus for Shock Wave Lithotripsy of Renal Stones
Brief Title: Efficacy and Safety of Narrow Focus (F1) Versus Wide Focus (F3) of Shock Wave Lithotripsy (SWL) for Renal Calculi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Yasser A. Noureldin, Assistant Professor of Urology, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD 1-11-2020
Record Dates: First submitted 2021-02-03; First posted 2021-02-18 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Renal Stone; Treatment Side Effects
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 will undergo Shock Wave Lithotripsy (SWL) with focal size 2mm (F1), and 3000 shocks
  Interventions: Procedure: Shock Wave Lithotripsy (SWL)
- Group 2 (Active Comparator): Group 2 will undergo Shock Wave Lithotripsy (SWL) with focal size 8mm (F3), and 3000 shocks
  Interventions: Procedure: Shock Wave Lithotripsy (SWL)

INTERVENTIONS:
Procedure: Shock Wave Lithotripsy (SWL) — Shock Wave Lithotripsy (SWL) with focal size 2mm (F1), and 3000 shocks or Shock Wave Lithotripsy (SWL) with focal size 8mm (F3), and 3000 shocks

SUMMARY:
This study aims to compare the narrow focus (F1) versus the wide focus (F3) in terms of the efficacy of Shock Wave Lithotripsy (SWL) in the management of renal calculi 1-2 cm and their injurious effect on the kidney.

DETAILED DESCRIPTION:
Recently, some Shock Wave Lithotripsy (SWL) devices have been announced in the market with a different focus points. One early experimental study found that stone disintegration is better with small focusing points than larger focusing points. Nevertheless, these findings, in terms of the efficacy of stone disintegration, need to be validated in-vivo. Furthermore, the effect of focal size on renal injury during SWL need to be studied as well. Therefore, the objectives of this study are to compare the effect of using the narrow focus of 2mm (F1) versus the wide focus of 8 mm (F3) on the Stone Free Rate (SFR) following SWL for renal stones 1-2cm and estimating renal injury effect of F1 vs. F3 by urinary renal injury markers such as neutrophil gelatinase-associated lipocalin (NGAL) for assessment of proximal and distal renal tubules injury & Kidney Injury Molecule-1 (KIM-1) for assessment of proximal renal tubules injury).

The SWL device:

Lithotripter type: Piezo Lith3000 plus ( from Richard Wolf, Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18years old) with 1-2 cm single renal stone.
2. Normal functioning kidney.

Exclusion Criteria:

1. Pregnancy.
2. Bleeding diatheses.
3. Radiolucent stones.
4. Radio-opaque stones with Hounsfield Unit (HU) > 1200
5. Patients with a pacemaker.
6. Active Urinary Tract Infection (UTI).
7. Severe skeletal malformations.
8. Morbid obesity with Body Mass Index (BMI) ≥40 kg/m2.
9. Renal artery aneurysm at the same site of the stone.
10. Anatomical obstruction distal to the stone.
11. Patients with renal impairment with serum creatinine > 1.2 mg/dL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy of Shock Wave Lithotripsy (SWL) by calculation of the percentage (%) of stone free | 1 year
  Assessment of efficacy of Shock Wave Lithotripsy (SWL) and its success by calculation of stone free (%) following each session with a maximum of 3 Shock Wave Lithotripsy (SWL) sessions, 2 weeks a part, using pelvi-abdominal Ultrasound (US) and Kidney-Ureter-Bladder (KUB) and the presence of significant residual stone >4 mm will be considered "non-stone free" and the final stone free status (%) will be calculated at one month following the last session of Shock Wave Lithotripsy (SWL).
  Shock Wave Lithotripsy (SWL) failure will be defined as failure to reach stone free status (%) one month after 3rd session.

SECONDARY OUTCOMES:
Assessment of the degree of renal injury using renal injury markers | 1 year
  Assessment of the degree of renal injury using renal injury markers as follow:
  - Urine analysis for neutrophil gelatinase-associated lipocalin (NGAL) (ng/dL) & Kidney Injury Molecule 1 (KIM-1) (ng/dL) will be measured measured with enzyme-linked immunosorbent assay (ELISA) method before, 2 hours after and 72 hours after the 1st Shock Wave Lithotripsy (SWL) session.
Assessment of the presence of peri-renal hematoma | 1 year
  Assessment of the presence of peri-renal hematoma will be conducted as follow:
  - Ultrasonography (US) will be done 24 hours after Shock Wave Lithotripsy (SWL) session to search for the presence of peri-renal hematoma and measure its size (cc).
Assessment of the changes in renal cortical thickness | 1 year
  Changes in the renal cortical thickness will be assessed as follow:
  - Ultrasonography (US) will be done before and after 6 months post Shock Wave Lithotripsy (SWL) for assessment of renal cortical thickness (mm) and the pre- and post-SWL measurements will be compared
Measurement of the changes in the Renal Resistive Index (RRI) | 1 year
  Renal Resistive Index (RRI) will be measured in the arcuate arteries using the following formula "RRI can be calculated as (peak systolic velocity - end diastolic velocity)/peak systolic velocity" before and 24 hours after Shock Wave Lithotripsy (SWL) using Doppler Ultrasound and changes will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Noureldin, MD, PhD, Principal Investigator — Benha University; Ahmed Abdelbaky, MD, PhD, Study Chair — Benha University; Walid Ibrahim, MD, PhD, Study Director — Benha University; Ezzat Elnahife, MD, Study Director — Benha University; Salah El Hamshary, MD, PhD, Study Director — Benha University
Locations (1):
- Faculty of Medicine, Benha University, Banhā, Kalyobiya, Egypt

REFERENCES:
- [Background] Turney BW, Reynard JM, Noble JG, Keoghane SR. Trends in urological stone disease. BJU Int. 2012 Apr;109(7):1082-7. doi: 10.1111/j.1464-410X.2011.10495.x. Epub 2011 Aug 26. PMID 21883851
- [Background] Connors BA, Evan AP, Blomgren PM, Handa RK, Willis LR, Gao S. Effect of initial shock wave voltage on shock wave lithotripsy-induced lesion size during step-wise voltage ramping. BJU Int. 2009 Jan;103(1):104-7. doi: 10.1111/j.1464-410X.2008.07922.x. Epub 2008 Aug 1. PMID 18680494
- [Background] Devarajan P. Biomarkers for the early detection of acute kidney injury. Curr Opin Pediatr. 2011 Apr;23(2):194-200. doi: 10.1097/MOP.0b013e328343f4dd. PMID 21252674
- [Background] Veser J, Jahrreiss V, Seitz C, Ozsoy M. The effect of focus size and intensity on stone fragmentation in SWL on a piezoelectric lithotripter. World J Urol. 2020 Oct;38(10):2645-2650. doi: 10.1007/s00345-019-03069-y. Epub 2020 Jan 10. PMID 31925550